CLINICAL TRIAL: NCT07307391
Title: Physiological Responses in Semi-professional Athletes: a Comparison of the Effects of Hot Weather Conditions
Brief Title: Exercise in Extreme Hot Weather Conditions
Acronym: EXHOTCON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Diego Fernández Lázaro, Professor Doctor, University of Valladolid
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025.14.11
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Heat Acclimation and Thermotolerance; Heat Effect
Keywords: Heat Stress; Exposure time; Gender difference; WBGT
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: A factorial experimental interventional study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- hot wet high (HWH) (Experimental): Air Temperature (ºC) 30.6±1.2 Relative Humidity (%) 68.6±1.3 Vapour Pressure (kPa) 1011±1.1 Bruel and Kjear (WBGT ºC) 27.3±0.8 Heat Stress (WBGT ºC) 27.8±0.8 Air Velocity (m/s) 0.45±0.19
  Interventions: Other: hot wet high (HWH)
- hot dry high (HDH) (Experimental): Relative Humidity (%) 39.7±0.3 Vapor Pressure (kPa) 29.0±1.2 Bruel and Kjear (WBGT ºC) 1007.9± 6.4 Heat Stress (WBGT ºC) 28.9±0.6 Air Velocity (m/s) 28.4±0.3
  Interventions: Other: hot dry high (HDH)
- hot dry low (HWL) (Experimental): Relative Humidity (%) 31.1±0.1 Vapor Pressure (kPa )67.1±1.0 Bruel and Kjear (WBGT ºC)1005.7±8.0 Heat Stress (WBGT ºC) 27.4±0.6 Air Velocity (m/s) 27.9±0.3
  Interventions: Other: Experimental: hot dry low (HWL)
- hot wet low (HWL) (Experimental): Relative Humidity (%) 39.8±0.1 Vapor Pressure (kPa) 26.4±0.4 Bruel and Kjear (WBGT ºC) 1004.7±10.7 Heat Stress (WBGT ºC) 28.3±0.3 Air Velocity (m/s) 27.7±0.1
  Interventions: Other: Experimental: hot wet low (HWL)

INTERVENTIONS:
Other: hot wet high (HWH) — Air Temperature (ºC) 30.6±1.2 Relative Humidity (%) 68.6±1.3 Vapour Pressure (kPa) 1011±1.1 Bruel and Kjear (WBGT ºC) 27.3±0.8 Heat Stress (WBGT ºC) 27.8±0.8 Air Velocity (m/s) 0.45±0.19
  Arms: hot wet high (HWH)
Other: hot dry high (HDH) — Relative Humidity (%) 39.7±0.3 Vapor Pressure (kPa) 29.0±1.2 Bruel and Kjear (WBGT ºC) 1007.9± 6.4 Heat Stress (WBGT ºC) 28.9±0.6 Air Velocity (m/s) 28.4±0.3
  Arms: hot dry high (HDH)
Other: Experimental: hot dry low (HWL) — Relative Humidity (%) 31.1±0.1 Vapor Pressure (kPa )67.1±1.0 Bruel and Kjear (WBGT ºC)1005.7±8.0 Heat Stress (WBGT ºC) 27.4±0.6 Air Velocity (m/s) 27.9±0.3
  Arms: hot dry low (HWL)
Other: Experimental: hot wet low (HWL) — Relative Humidity (%) 39.8±0.1 Vapor Pressure (kPa) 26.4±0.4 Bruel and Kjear (WBGT ºC) 1004.7±10.7 Heat Stress (WBGT ºC) 28.3±0.3 Air Velocity (m/s) 27.7±0.1
  Arms: hot wet low (HWL)

SUMMARY:
Background: Core body temperature increases in hot climates due to exercise workload, disrupting heat gain and loss of balance. The human thermoregulatory system regulates core body temperature through factors such as metabolic heat production, air temperature, humidity, and clothing. The study investigates physiological thermoregulatory responses in semiprofessional athletes during walking and jogging in different climatic conditions.

Methods: A factorial experimental interventional design was used to evaluate different physical activity (low (L)=5 km/h and high (H)=8 km/h) and climatic conditions within the Thermal Environment Laboratory at Lund University, Sweden. The temperature within the climatic chamber was set at 40°C and 31°C, with a relative humidity of 20% and 70%, (hot dry (HD) and hot humid (HW), respectively, to account for a 28°C WBGT. The study used independent T-tests, ANOVA and simple linear regression models to analyse the physiological responses of semiprofessional athletes under different test conditions, comparing gender differences.

ELIGIBILITY:
Inclusion Criteria:

* Participation at the regional competition level
* Receiving monetary remuneration for their sports engagement
* Participating in sports activities in the previous six years
* Average training experience of 6.0±1.4 years
* A weekly volume of 6.3±0.7 days for 2.3±0.7 hours (h)·day-¹.

Exclusion Criteria:

* A 2 kg weight change in the previous month
* Adherence to special diets
* Use of nutritional supplements
* Smoking
* An acute or chronic communicable or noncommunicable disease
* Heat allergic problems.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Exposure Time | Just one day, the day of the test, in those weather conditions
  duration an athlete is exposed to a specific intensity or environmental condition
Heart Rate | Just one day, the day of the test, in those weather conditions
  measures how hard your heart works to gauge fitness
Oxygen Uptake | Just one day, the day of the test, in those weather conditions
  how much oxygen your body uses during activity

SECONDARY OUTCOMES:
Core Body Temperature | Just one day, the day of the test, in those weather conditions
  the body's internal temperature regulation
Skin Temperature | Just one day, the day of the test, in those weather conditions
  The temperature of your body's surface
Body Temperature | Just one day, the day of the test, in those weather conditions
  the internal heat level of the human body
Sweat Rate | Just one day, the day of the test, in those weather conditions
  the amount of fluid your body loses through sweat per hour during exercise
Perceived Exertion Level | Just one day, the day of the test, in those weather conditions
  is a subjective scale that measures how hard your body feels it's working during exercise
Thermal Sensation Level | Just one day, the day of the test, in those weather conditions
  The Thermal Sensation Level is a standardized, subjective rating system used to quantify a person's perception of warmth or coolness in their environment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, University of Valladolid Soria Campus, Soria, Soria 42004, Soria, Soria, Spain